CLINICAL TRIAL: NCT06874244
Title: Randomized Prospective Split Mouth Clinical Evaluation of no Needle Dental Anesthesia Compared to Syringe Anesthesia Delivery
Brief Title: Clinical Evaluation of no Needle Dental Anesthesia Compared to Syringe Anesthesia Delivery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: Henley Ion (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 4944
Record Dates: First submitted 2025-03-03; First posted 2025-03-13 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-06

CONDITIONS: Local Anesthesia Injection Pain
Keywords: Local Anesthesia
MeSH Terms: interventions — Anesthesia, Local; Lidocaine; Oxymetazoline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Iontophoresis of Tetracaine and oxymetazoline (Experimental)
  Interventions: Drug: Iontophoresis of Tetracaine and oxymetazoline
- Local Anesthesia (lidocaine hydrochloride) (Active Comparator)
  Interventions: Drug: Local Anesthesia (lidocaine hydrochloride)

INTERVENTIONS:
Drug: Local Anesthesia (lidocaine hydrochloride) — Injection of lidocaine as local anesthesia
  Arms: Local Anesthesia (lidocaine hydrochloride)
Drug: Iontophoresis of Tetracaine and oxymetazoline — Injecting Tetracaine Hydrochloride 4% with 0.5% Oxymetazoline to the oral tissue using iontophoresis technique
  Arms: Iontophoresis of Tetracaine and oxymetazoline

SUMMARY:
The purpose of the study is to evaluate two different ways to administer the numbing solution. One is with a conventional needle and syringe the other method iontophoresis is a machine that supplies a weak current through electrodes that touch your teeth. Both methods use an anesthesia solution to make your teeth numb but the iontophoresis system contains no needle and the delivery device does not penetrate the gum.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age at the time of consent

Subject is able to provide their own informed consent

Subject has a minimum 24 teeth/subject and 6 teeth per quadrant

Subject has an Approximal Plaque Index score ≤ 40% as assessed via explorer and without the use of plaque-disclosing agents

Subject must be able to speak and understand English

Subject is able and willing to return for all scheduled study visits

Subject to able to make dental appointments

Subject should not be a pregnant female

Subject meets the Level-I or Level-II classification criteria of the American

Society of Anesthesiologists (ASA) Physical Status Classification System For Dental Patient Care

Exclusion Criteria:

* Subject has any of the following:

  * rampant caries
  * chronic periodontitis
  * salivary gland dysfunction

Subject is unable, for any reason, to tolerate the procedure time required to place the restorations

Subject has unacceptable oral hygiene (e.g., chronic moderate to heavy plaque accumulation along the gumline)

Subject is planned to be enrolled in another investigational trial that requires additional interventions at any time during the study

Subject is using a whitening agent at any time during this study.

Subject has history of allergic reaction to anesthetic medications

Subject with uncontrolled systemic disease or conditions

Subject is having acute or chronic myofascial pain or neuropathic conditions

Subject taking long-term analgesics for their systemic conditions

Subject presenting with acute dental pain

Subject requiring IV sedation or nitrous oxide sedation or oral sedation for anxiety

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Pain response in the gingiva | Up to 1 hour
  Pain response in the gingiva will be recorded as a yes/no after a painful stimulus is applied using a probe on the buccal and palatal soft tissues.
Cold pulp test | Up to 1 hour
  The pulpal response will be assessed using a cold pulp test as yes/ no response.

SECONDARY OUTCOMES:
Pain scale: Visual analog scale | Baseline and 2 minutes after delivery of anesthesia.
Beck's anxiety scale | Baseline and 2 minutes after delivery of anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- LSUHSC School of Dentistry, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No